CLINICAL TRIAL: NCT03405896
Title: The Validity and Reliability of a Wearable System for Assessing Turning Characteristics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YM106038E
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Ambulation Difficulty
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal subjects (Experimental)
  Interventions: Other: Turning

INTERVENTIONS:
Other: Turning — start to walk with normal speed, and then turn to approach the terminal under different angle.

SUMMARY:
The Validity and Reliability of a Wearable System for Assessing Turning Characteristics.

DETAILED DESCRIPTION:
Subjects are reclaimed to finish several turning task under different turning angle.

The wearable system is patched on both subjects' legs and waist, to assess turning characteristics under different turning angle.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 10 m independently without any device.

Exclusion Criteria:

* Dizzy causing by eye disorders or vestibular disease.
* Any disease which involved in gait performance.
* Can't follow the order by investigator during task.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-08-23 (Estimated); Study Completion 2019-08-23 (Estimated)

PRIMARY OUTCOMES:
Turning step count | pre-test and post-test within a week
  record numbers of step during turning
Turing time | pre-test and post-test within a week
  record second which subject spend during turning
Stride length during turning | pre-test and post-test within a week
  record the distance of bipedal stride length respectively
Walking speed approached turning | pre-test and post-test within a week
  record the velocity and change of velocity before start turning
Turning angle | pre-test and post-test within a week
  record the total turning angle and bipedal turning angle each step

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan